CLINICAL TRIAL: NCT04676555
Title: Time and Motion Study for Ocrelizumab and Ofatumumab Administration in Relapsing Multiple Sclerosis
Acronym: TIMIOS
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: COMB157G2004
Record Dates: First submitted 2020-12-16; First posted 2020-12-21 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Relapsing Forms of Multiple Sclerosis
Keywords: Relapsing forms of Multiple Sclerosis; RMS; Ocrelizumab; Ofatumumab; TIMIOS
MeSH Terms: interventions — ocrelizumab; ofatumumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Ocrelizumab: Ocrelizumab is administered intravenously (IV) under the guidance of a specialized physician and followed by one-hour observation after the infusion. It requires a corticosteroid pre-medication and some antipyretics may also be administered.
  Interventions: Drug: Ocrelizumab
- Ofatumumab: Ofatumumab is administered through a subcutaneous injection and allows self-administration after training.
  Interventions: Drug: Ofatumumab

INTERVENTIONS:
Drug: Ocrelizumab — There is no treatment allocation. Patients administered Ocrelizumab by prescription that have started before inclusion of the patient into the study will be enrolled.
  Groups: Ocrelizumab
Drug: Ofatumumab — There is no treatment allocation. Patients administered Ofatumumab by prescription that have started before inclusion of the patient into the study will be enrolled.
  Groups: Ofatumumab

SUMMARY:
This is an observational cross-sectional study of Ocrelizumab or Ofatumumab administrations for Relapsing forms of Multiple Sclerosis (RMS) in selected sites in the US, the UK and Australia.

DETAILED DESCRIPTION:
Patients with RMS receiving Ocrelizumab or Ofatumumab will be recruited to measure the time spend for Healthcare Providers (HCP) (neurologist, nurse and hospital pharmacist) on preparing, administering the medication and following up with the patient.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of 18 or more years of age.
* Patients with confirmed diagnosis of RMS (CIS, RRMS or aSPMS) following 2017 McDonnald criteria.
* Patients currently prescribed with Ocrelizumab or Ofatumumab to treat MS according to the Summary of Product Characteristics (SmPC). The decision must be based on patient disease and taken before the decision of inviting the patient to participate in this study.
* Patients literate in English.
* Patients must provide informed consent to participate in the study.

Exclusion Criteria:

* Patients currently participating in any other RMS clinical trial.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed of RMS will be recruited if they have been prescribed either Ocrelizumab of Ofatumumab. The person accompanying the patient will be invited to participate as a caregiver.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2021-05-11 (Actual); Primary Completion 2021-10-21 (Actual); Study Completion 2021-10-21 (Actual)

PRIMARY OUTCOMES:
Time spent by Healthcare Providers (staff) in the preparation, administration and post-treatment observation of Ocrelizumab and Ofatumumab | Ocrelizumab: Initial dose (week 0), Loading dose (week 2), Subsequent dose (month 6, month 12, or month 18). Ofatumumab: Initial dose (week 0), Loading dose (week 1 or week 2), Subsequent dose (week 4, week 8, or week 12)
  Describe and compare the time spent by Healthcare Providers (in minutes) in the treatment preparation, administration and post-treatment observation of Ocrelizumab and Ofatumumab in patients with Relapsing forms of Multiple Sclerosis at each event (initial, loading and subsequent doses).

SECONDARY OUTCOMES:
Healthcare resources used, in terms of consumables in the treatment preparation and administration of Ocrelizumab and Ofatumumab | Ocrelizumab: Initial dose (week 0), Loading dose (week 2), Subsequent dose (month 6, month 12, or month 18). Ofatumumab: Initial dose (week 0), Loading dose (week 1 or week 2), Subsequent dose (week 4, week 8, or week 12)
  Describe and compare the healthcare resources used, in terms of number of consumables used, in the treatment preparation and administration of Ocrelizumab and Ofatumumab for RMS patients at each event.
Cost of staff and consumables used in the treatment preparation, administration and post-treatment observation of Ocrelizumab and Ofatumumab | Ocrelizumab: Initial dose (week 0), Loading dose (week 2), Subsequent dose (month 6, month 12, or month 18). Ofatumumab: Initial dose (week 0), Loading dose (week 1 or week 2), Subsequent dose (week 4, week 8, or week 12)
  Describe and compare the cost of staff and consumables used in the treatment preparation, administration and post-treatment observation of Ocrelizumab and Ofatumumab for RMS patients at each event.
Healthcare resources used, in terms of staff time in managing the adverse events occurred during the administration and post treatment observation of Ocrelizumab and Ofatumumab | Ocrelizumab: Initial dose (week 0), Loading dose (week 2), Subsequent dose (month 6, month 12, or month 18). Ofatumumab: Initial dose (week 0), Loading dose (week 1 or week 2), Subsequent dose (week 4, week 8, or week 12)
  Describe and compare the healthcare resources used, in terms of staff time in managing the adverse events occurred during the administration and post treatment observation of Ocrelizumab and Ofatumumab in RMS patients at each event.
Healthcare resources used, in terms of consumables in managing the adverse events occurred during the administration and post treatment observation of Ocrelizumab and Ofatumumab | Ocrelizumab: Initial dose (week 0), Loading dose (week 2), Subsequent dose (month 6, month 12, or month 18). Ofatumumab: Initial dose (week 0), Loading dose (week 1 or week 2), Subsequent dose (week 4, week 8, or week 12)
  Describe and compare the healthcare resources used, in terms of number of consumables used in managing the adverse events occurred during the administration and post treatment observation of Ocrelizumab and Ofatumumab in RMS patients at each event.
Indirect cost as assessed by the Work Productivity and Activity Impairment Questionnaire: Multiple sclerosis (WPAI:MS | Ocrelizumab: Initial dose (week 0), Loading dose (week 2), Subsequent dose (month 6, month 12, or month 18). Ofatumumab: Initial dose (week 0), Loading dose (week 1 or week 2), Subsequent dose (week 4, week 8, or week 12)
  Describe and compare as assessed by the Work Productivity and Activity Impairment Questionnaire: Multiple sclerosis (WPAI:MS) at each event.
  The WPAI measures four types of scores: 1. Absenteeism (work time missed); 2. Presenteeism (impairment at work / reduced on-the-job effectiveness); 3. Overall productivity loss (overall impairment / absenteeism plus presenteeism); 4. Usual activity Impairment. WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity
Indirect cost as assessed by the Work Productivity and Activity Impairment Questionnaire: Caregiver (WPAI:CG) | Ocrelizumab: Initial dose (week 0), Loading dose (week 2), Subsequent dose (month 6, month 12, or month 18). Ofatumumab: Initial dose (week 0), Loading dose (week 1 or week 2), Subsequent dose (week 4, week 8, or week 12)
  Describe and compare as assessed by the Work Productivity and Activity Impairment Questionnaire: Caregiver (WPAI:CG), at each event.
  The WPAI measures four types of scores: 1. Absenteeism (work time missed); 2. Presenteeism (impairment at work / reduced on-the-job effectiveness); 3. Overall productivity loss (overall impairment / absenteeism plus presenteeism); 4. Usual activity Impairment. WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Novartis Investigative Site, Lutherville, Maryland, United States
- Novartis Investigative Site, Parkville, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No